CLINICAL TRIAL: NCT02224378
Title: Prediction of Fluid Responsiveness in Atrial Fibrillation Patients Who Underwent Valvular Heart Surgery: Peep-induced Increase in Central Venous Pressure vs. Passive Leg Raising
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 4-2011-0686
Record Dates: First submitted 2014-08-19; First posted 2014-08-25 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2015-03

CONDITIONS: Valvular Heart Surgery
Keywords: fluid responsiveness; atrial fibrillation; passive leg raising; central venous pressure; valvular heart surgery
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- peep induced CVP (Experimental)
  Interventions: Procedure: peep induced CVP
- passive leg raising(PLR) (Active Comparator)
  Interventions: Procedure: passive leg raising(PLR)

INTERVENTIONS:
Procedure: peep induced CVP
  Arms: peep induced CVP
Procedure: passive leg raising(PLR)
  Arms: passive leg raising(PLR)

SUMMARY:
Dynamic indices of preload depending on the heart-lung interaction require sinus rhythm and cannot be applied to patients with atrial fibrillation. PEEP-induced increase in central venous pressure (CVP) was shown to be a valid predictor of fluid responsiveness after cardiac surgery in patients with sinus rhythm, and was speculated to be of value in patients with rhythm other than sinus. The aim of this study is to assess the predictability of PEEP-induced increase in CVP and passive leg raising (PLR)-induced changes in stroke volume index (SVI) on fluid responsiveness in patients with atrial fibrillation following valvular heart surgery.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥20
2. atrial fibrillation patients who underwent elective valvular heart surgery

Exclusion Criteria:

1. age < 20
2. LV ejection fraction < 40%
3. any pulmonary disease
4. end stage renal disease
5. high intrabdominal pressure patient
6. contraindication of passive leg raising
7. deep vein thrombosis

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2012-03; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
fluid responsiveness | 1hr after arriving at ICU
  1. ventilator peep setting was adjusted to 0cmH2O as baseline
  2. Then peep was increased to 10cmH2O for 5 min.
  3. We set peep to baseline 0cmH2O again, making patients to semirecumbent position following passive leg raising at 30 degree for 5 min.
  4. After that, 300 ml of hydroxyethyl starch 130/0.4 was infused in the supine position for 10-20 min and haemodynamic variables including SVI were assessed 5 min after completion of fluid challenge.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology & Pain Medicine, Yonsei university college of medicine, Seoul, Seoul, South Korea